CLINICAL TRIAL: NCT02390973
Title: Surgery Versus Best Medical Management for the Long Term Remission of Type 2 Diabetes and Related Diseases (REMISSION)
Acronym: REMISSION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Johnson & Johnson Medical Products (Unknown); Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Laurent Biertho, Principal Investigator, Laval University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Remission
Record Dates: First submitted 2015-02-16; First posted 2015-03-18 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Bariatric Surgery Candidate; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Gastric Bypass; Biliopancreatic Diversion; Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sleeve gastrectomy (Active Comparator)
  Interventions: Procedure: Sleeve Gastrectomy
- Roux-en-Y Gastric Bypass (Active Comparator)
  Interventions: Procedure: Roux-en-Y Gastric Bypass
- Biliopancreatic Diversion (Active Comparator)
  Interventions: Procedure: Biliopancreatic Diversion with Duodenal Switch
- Control (Active Comparator): the best medical management of their diabetes, non-surgical group
  Interventions: Other: Medical management

INTERVENTIONS:
Procedure: Sleeve Gastrectomy
  Arms: Sleeve gastrectomy
Procedure: Roux-en-Y Gastric Bypass
  Arms: Roux-en-Y Gastric Bypass
Procedure: Biliopancreatic Diversion with Duodenal Switch
  Arms: Biliopancreatic Diversion
Other: Medical management
  Arms: Control

SUMMARY:
Bariatric surgery procedures induce weight loss through restriction and/or malabsorption. The mechanisms underlying type 2 diabetes remission and others metabolic improvements after Roux-en-Y Gastric Bypass (RYGB), sleeve gastrectomy (SG) or biliopancreatic diversion with duodenal switch (BPD-DS) have not yet been formally studied. The investigators propose a longitudinal study with the overall objective of measuring the long-term impact of these three bariatric surgeries (RYGB, SG, BPD-DS) on metabolic, renal and cardiovascular fate in patients with type 2 diabetes. The investigators overall hypothesis is that some bariatric procedures generate hitherto unrecognized effects on many disease-related outcomes, which greatly contributes to their beneficial impact in diabetic patients. The investigators propose 3 specific aims: 1) to establish the long term effect of the three surgeries on the metabolic recovery and quality of life in groups of diabetic patients treated with insulin, hypoglycemic agents or diet; 2) to establish the long term impact of the three surgeries on renal and cardiovascular functions in subgroup of patients with these conditions; 3) to compare metabolic impact of surgeries to those of best medical care for diabetes in a non-surgical control group. For most severely obese patients, lifestyle interventions, perhaps effective in inducing short-lived weight losses, are ineffective for long-term weight loss maintenance and durable metabolic recovery. The increasing popularity of obesity surgeries calls for a better understanding of the underlying mechanisms. This is especially true and urgent when considering that knowledge on the relative impact of each procedure (i.e. SG vs. RYGB and BPD-DS) in resolving T2D is still limited. Better knowledge on each of the procedures will allow stronger scientific rationale for selecting the right surgery for the right patient and improve care for the severely obese individual.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35
* type 2 diabetes
* HbA1c ≥ 6,5 % or fasting glycemia ≥7mmol/l or non-fasting glycemia ≥11mmol/l
* able to consent

Exclusion Criteria:

* pregnancy
* past esophageal, gastric or bariatric surgery
* irritable bowel, unexplained intermittent vomiting, severe abdominal pain, chronic diarrhea or constipation
* history of gastric or duodenal ulcers
* pre-operatory hypoalbuminemy
* history of renal, hepatic, cardiac or pulmonary severe disease
* taken of corticosteroid in the last month
* evidence of psycological problem that may affect the capacity to understand the project and to comply with the medical recommandations
* history of drug use or alcool abuse in the last 12 months
* history of gastro-intestinal inflammatory diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 408 (Estimated)
Dates: Start 2015-03; Primary Completion 2027-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Type 2 diabetes remission rate | from baseline up to 60 months
  percent of patient achieving type 2 diabetes remission in each groups

SECONDARY OUTCOMES:
Change in microalbuminuria | from baseline up to 60 months
  Normalisation of A/C ratio after surgery
Change in retinopathy | from baseline up to 60 months
Hypertension remission rate | from baseline up yo 60 months
  percent of patient achieving hypertension remission in each groups
GERD remission rate | from baseline up to 60 months
  percent of patient achieving gastro-esophageal reflux disease resolution in each groups
Quality of life | from baseline up to 60 months
  quality of life after surgery eveluated with questionnaires
Sleep apnea remission rate | from baseline up to 60 months
  percent of patient achieving sleep apnea remission in each groups
weight loss | from baseline up to 60 months
  weight loss (kg)
Regression of liver disease | from baseline up to 60 months
  regression of liver disease documented by percutaneous liver biopsy after surgery
Dislipidemia remission | from baseline up to 60 months
  percent of patient achieving dislipidemia remission in each groups

OTHER OUTCOMES:
short-term complications | baseline up to 4 month
  comparaison of intra-operative, post-operative and in-hospital complications between groups using clavien classification
Long-term complications | baseline up to 60 months
  Vital status and long-term complications including cardiovascular events, micro- or macro-vascular complications, cancer, psychiatric events, bone fractures, operations, readmission related or unrelated to the surgery, changes in medical treatment will be compared between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Bouchard-Mercier A, de Toro-Martin J, Nadeau M, Lescelleur O, Lebel S, Richard D, Biertho L, Tchernof A, Vohl MC. Molecular remodeling of adipose tissue is associated with metabolic recovery after weight loss surgery. J Transl Med. 2022 Jun 23;20(1):283. doi: 10.1186/s12967-022-03485-6. PMID 35739539
- [Derived] Carreau AM, Noll C, Blondin DP, Frisch F, Nadeau M, Pelletier M, Phoenix S, Cunnane SC, Guerin B, Turcotte EE, Lebel S, Biertho L, Tchernof A, Carpentier AC. Bariatric Surgery Rapidly Decreases Cardiac Dietary Fatty Acid Partitioning and Hepatic Insulin Resistance Through Increased Intra-abdominal Adipose Tissue Storage and Reduced Spillover in Type 2 Diabetes. Diabetes. 2020 Apr;69(4):567-577. doi: 10.2337/db19-0773. Epub 2020 Jan 8. PMID 31915151